CLINICAL TRIAL: NCT01117623
Title: Open Label, Phase I Study to Determine the Safety, Tolerability, Maximum Tolerated Dose, Pharmacokinetics, and Biomarker Status of BAY73-4506 in Patients With Advanced Malignancies
Brief Title: Continuous Dosing of BAY73-4506 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 11651
Record Dates: First submitted 2010-02-11; First posted 2010-05-05 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Neoplasm
Keywords: Oncology patients with advanced disease; BAY73-4506
MeSH Terms: conditions — Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Arm 1 (Experimental)
  Interventions: Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg
- Arm 2 (Experimental)
  Interventions: Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg
- Arm 3 (Experimental)
  Interventions: Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg
- Arm 4 (Experimental)
  Interventions: Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg
- Arm 5 (Experimental)
  Interventions: Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg
- Arm 6 (Experimental)
  Interventions: Drug: HCC Child-Pugh A expansion cohort: Regorafenib 100 mg
- Arm 7 (Experimental)
  Interventions: Drug: HCC Child-Pugh B expansion cohort: Regorafenib 100 mg
- Arm 8 (Experimental)
  Interventions: Drug: NSCLC expansion cohort: Regorafenib 100 mg

INTERVENTIONS:
Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg — Participants in the dose-escalation cohort received a single 20 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral co-precipitate (CP) tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 1
Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg — Participants in the dose-escalation cohort received a single 40 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 40 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 2
Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg — Participants in the dose-escalation cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 3
Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg — Participants in the dose-escalation cohort received a single 120 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 120 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 4
Drug: Escalation cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg — Participants in the dose-escalation cohort received a single 140 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 140 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 5
Drug: HCC Child-Pugh A expansion cohort: Regorafenib 100 mg — Hepatocellular carcinoma (HCC) Participants with Child Pugh A in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 6
Drug: HCC Child-Pugh B expansion cohort: Regorafenib 100 mg — Hepatocellular carcinoma (HCC) Participants with Child Pugh B in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 7
Drug: NSCLC expansion cohort: Regorafenib 100 mg — Non-small cell lung cancer (NSCLC) participants in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
  Arms: Arm 8

SUMMARY:
Continuous dosing of BAY73-4506 in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Patients with advanced, histologically or cytologically confirmed solid tumors, malignant lymphomas, or multiple myeloma refractory to any standard therapy
* Radiographical, hematological or clinically evaluable tumor
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements:

  * Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* History of cardiac disease: congestive heart failure (CHF) > New York Heart Association (NYHA) Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months or unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management
* History of HIV infection or chronic hepatitis B or C
* Active clinically serious infections (> Grade 2 NCI Common Terminology Criteria for Adverse Events v3.0)
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 2 weeks prior to study entry and is clinically stable with respect to the tumor at the time of study entry. Patients with brain metastases must not be undergoing acute steroid therapy or steroid taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* Substance abuse, medical, psychological or social conditions that may interfere with the patient178s participation in the study or evaluation of the study results
* Radiotherapy to the target lesions within 3 weeks prior to Day 1, Cycle 1 (first dose of study drug). (Palliative radiotherapy will be allowed). Radiotherapy to the target lesions during study will be regarded as progressive disease
* Previous or concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis and T1] or any cancer curatively treated > 3 years prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - Los Angeles, California
  - Aurora, Colorado
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with advanced, histologically or cytologically confirmed solid tumors (including non-small-cell lung cancer (NSCLC) participants enrolled in the expansion portion of the study), malignant lymphomas, or multiple myeloma were enrolled in 5 centers in the USA from 01 FEB 2007 to 22 Apr 2011.
Pre-assignment Details: 109 (73 male and 36 female) participants were screened according to the inclusion and exclusion criteria to determine their appropriateness for inclusion in the study, and 86 (54 male and 32 female) participants were included at 5 centers, valid for safety population, 81 participants valid for ITT efficacy analysis and PK population.
Groups:
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg: Participants in the dose-escalation cohort received a single 20 mg oral co-precipitate (CP) tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
Period: Overall Study
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Started | 3 | 8 | 11 | 6 | 10 | 16 | 6 | 26
ITT Efficacy Analysis Population | 3 | 8 | 11 | 5 | 10 | 16 | 6 | 22
PK Population | 3 | 8 | 10 | 6 | 10 | 14 | 6 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 11 | 6 | 10 | 16 | 6 | 26
Not completed — Adverse Event | 0 | 2 | 4 | 0 | 2 | 0 | 0 | 2
Not completed — Disease progression, recurrence, relapse | 3 | 6 | 5 | 6 | 8 | 14 | 5 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Not completed — Non-compliance with study medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Invest. text: completed all planned txs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg: Participants in the dose-escalation cohort received a single 20 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg: Participants in the dose-escalation cohort received a single 40 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg: Participants in the dose-escalation cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg: Participants in the dose-escalation cohort received a single 120 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg: Participants in the dose-escalation cohort received a single 140 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg: Hepatocellular carcinoma (HCC) Participants with Child Pugh A status in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg: Hepatocellular carcinoma (HCC) Participants with Child Pugh B status in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg | Total
Number analyzed (Participants) | 3 | 8 | 11 | 6 | 10 | 16 | 6 | 26 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (8.1) | 55.3 (13.1) | 61.9 (8.8) | 59.2 (10.7) | 55.7 (13.7) | 56.6 (13.2) | 56.7 (13.1) | 62.4 (12.2) | 59.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 4 | 3 | 7 | 4 | 2 | 9 | 32
  Male | 3 | 5 | 7 | 3 | 3 | 12 | 4 | 17 | 54

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose level, which could be given to 6 participants such that no more than 1 participant (less than 33%) experienced a dose-limiting toxicity (DLT).
Time Frame: Within first 4 weeks of treatment
Population: Safety Population; dose escalation cohorts only
Measure: Number; unit: mg
Groups:
- Regorafenib, 20 mg, 40 mg, 100 mg, 120 mg, 140 mg: Participants in the dose-escalation cohort received a single 20 mg, 40 mg, 100 mg, 120 mg, 140 mg oral CP tablet of regorafenib respectively on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 20 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
Arm/Group | Regorafenib, 20 mg, 40 mg, 100 mg, 120 mg, 140 mg
Number analyzed (Participants) | 37
mg | 100

2. Primary Outcome: Maximum Observed Plasma Concentration After Single Dose Administration (Cmax)
Description: Cmax refers to the highest measured drug concentration, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: Blood samples were collected on Cycle 1, Day 1. Samples were drawn at the following time points: 0 h pre-dose, 0.5, 1, 2, 4, 8, 10, 24, and 48 h post-dose
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmax in at least one analyte was 1 (M5) in 20mg; 7 (regorafenib and M2) and 5 (M5) in 40mg; 13 (M5) in HCC Child-Pugh A; 22 (M5) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
mg/L
  Regorafenib (n=3,7,10,6,10,14,4,24) | 0.330 (14.8) | 0.422 (27.4) | 1.25 (30.7) | 1.87 (24.0) | 1.90 (51.2) | 1.38 (98) | 1.42 (76) | 1.25 (68.5)
  M2 (BAY75-7495) (n=3,7,10,6,10,14,4,24) | 0.0181 (244) | 0.0867 (110) | 0.401 (51.2) | 0.645 (43.2) | 0.606 (97.2) | 0.42 (154) | 0.54 (129) | 0.388 (190)
  M5 (BAY81-8752) (n=1,5,10,6,10,13,4,22) | 0.00290 (NA) — we have one data point only, n=1, calculation not possible | 0.00738 (124) | 0.0299 (118) | 0.0459 (59.2) | 0.0500 (140) | 0.036 (110) | 0.035 (352) | 0.321 (142)

3. Primary Outcome: Area Under the Concentration vs. Time Curve From Zero to Infinity After Single (First) Dose (AUC)
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 2
Population: PK population; Number of Participants with at least one evaluable AUC were 5 (regorafenib) and 6 (M2) in 40mg; 5 (regorafenib and M2) in 100 mg; 3 (M2) in 120 mg; 6 (regorafenib and M2) in 140 mg; 9 (regorafenib), 10 (M2) and 1 (M5) in HCC Child Pugh A; 3 (regorafenib) and 2 (M2) in HCC Child Pugh B; 19 (regorafenib) and 16 (M2) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
mg*h/L
  Regorafenib (n=3,5,5,6,6,9,3,19) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 16.3 (76.3) | 43.7 (34.9) | 52.9 (64.6) | 52.5 (66.4) | 45.2 (84.3) | 57.7 (30.9) | 33.5 (43.9)
  M2 (BAY75-7495) (n=3,6,5,3,6,10,2,16) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 3.53 (161) | 12.8 (37.0) | 21.0 (71.5) | 19.5 (20.3) | 15.3 (69.9) | 27.2 (74.6) | 11.6 (77.8)
  M5 (BAY81-8752) (n=3,8,10,6,10,1,4,24) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 15.8 (NA) — we have one data point only, n=1, calculation not possible | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations)

4. Primary Outcome: Cmax at Steady State During a Dosing Interval (Cmax,ss)
Description: Cmax,ss refers to the highest measured drug concentration, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample, after multiple dose administration and after a steady state concentration has been reached.
Time Frame: Blood samples were collected at on Cycle 2, Day 1 and on Cycle 3, Day 1 for expansion cohort. Samples were drawn at the following time points: 0 h pre-dose, 0.5, 1, 2, 4, 8, 10 and 24h post-dose.
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmax,ss in at least one analyte were 6 in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
mg/L
  Regorafenib (n=3,6,6,2,3,0,1,5) | 1.27 (19.4) | 1.50 (37.0) | 4.27 (22.9) | 3.62 (5.77) | 5.37 (30.9) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 2.69 (NA) — we have one data point only, n=1, calculation not possible | 2.55 (92.4)
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 0.0912 (39.5) | 0.520 (74.3) | 2.48 (36.3) | 2.97 (217) | 2.20 (106) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 2.40 (NA) — we have one data point only, n=1, calculation not possible | 0.911 (126)
  M5 (BAY81-8752) (n=3,6,6,2,3,0,1,5) | 0.00911 (15.7) | 0.174 (151) | 1.38 (87.0) | 3.29 (1400) | 0.948 (343) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 1.59 (NA) — we have one data point only, n=1, calculation not possible | 0.349 (153)

5. Primary Outcome: AUC From Time 0 to 24 Hours at Steady State(AUC(0-24),ss)
Description: AUC(0-24),ss is a measure of systemic drug exposure over 24 hours, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample, after multiple dose administration and after a steady state concentration has been reached.
Time Frame: Blood samples were collected on Cycle 2, Day 1 and on Cycle 3, Day 1 for expansion cohort. Samples were drawn at the following time points: 0 h pre-dose, 0.5, 1, 2, 4, 8, 10 and 24h post-dose.
Population: Pharmacokinetic population; Number of Participants with an evaluable AUC(0-24),ss in at least one analyte in at least one analyte were 6 in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
mg*h/mL
  Regorafenib (n=3,6,6,2,3,0,1,5) | 12.9 (21.2) | 18.1 (35.9) | 49.6 (18.5) | 40.6 (32.9) | 60.4 (18.5) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 39.2 (NA) — we have one data point only, n=1, calculation not possible | 35.8 (83.9)
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 1.11 (42.9) | 7.20 (56.7) | 31.5 (25.2) | 40.9 (245) | 29.7 (88.8) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 46.8 (NA) — we have one data point only, n=1, calculation not possible | 14.6 (104)
  M5 (BAY81-8752) (n=3,6,6,2,3,0,1,5) | 0.122 (18.7) | 2.22 (136) | 18.6 (58.1) | 44.4 (3050) | 12.9 (231) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 34.3 (NA) — we have one data point only, n=1, calculation not possible | 6.17 (133)

6. Secondary Outcome: AUC From Time 0 to the Last Data Point > Lower Limit of Quantification (LLOQ) (AUC(0-tlast))
Description: The AUC(0-tlast) is a measure of systemic drug exposure from time 0 up to the time point at which the last measurable drug could be detectable, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: as for outcome 2
Population: Pharmacokinetic population; Number of Participants with an evaluable AUC(0-tlast) in at least one analyte were 1(M-5) in 20mg; 7 (regorafenib and M-2) and 5 (M-5) in 40mg; 13 (M-5) in HCC Child Pugh A; 22 (M5) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
mg*h/L
  Regorafenib (n=3,7,10,6,10,14,4,24) | 7.98 (28.0) | 9.12 (38.8) | 32.7 (37.9) | 33.5 (60.4) | 35.8 (57.0) | 26.8 (67.5) | 33.0 (112) | 18.7 (55.3)
  M2 (BAY75-7495) (n=3,7,10,6,10,14,4,24) | 0.384 (330) | 2.02 (108) | 11.3 (47.4) | 14.2 (53.4) | 13.6 (82.6) | 8.84 (122) | 13.4 (194) | 6.54 (156)
  M5 (BAY81-8752) (n=1,5,10,6,10,13,4,22) | 0.0275 (NA) — we have one data point only, n=1, calculation not possible | 0.165 (254) | 0.976 (111) | 1.51 (71.1) | 1.54 (71.1) | 1.02 (122) | 0.821 (587) | 0.821 (254)

7. Secondary Outcome: Area Under the Concentration vs. Time Curve From Zero to Infinity After Single (First) Dose Divided by Dose (AUC/D)
Description: The AUC/D is a measure of systemic drug exposure (AUC) after the first single dose, which is then divided by that dose. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 2
Population: PK population; Number of Participants with at least one evaluable AUC/D were 5 (regorafenib) and 6 (M-2) in 40mg; 5 (regorafenib and M-2) in 100 mg; 3 (M-2) in 120 mg; 6 (regorafenib and M-2) in 140 mg; 9 (regorafenib), 10 (M-2) and 1 (M5) in HCC Child Pugh A; 3 (regorafenib) and 2 (M-2) in HCC Child Pugh B; 19 (regorafenib) and 16 (M-2) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
h/L
  Regorafenib (n=3,5,5,6,6,9,3,19) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 0.407 (76.3) | 0.437 (34.9) | 0.441 (64.6) | 0.375 (66.4) | 0.452 (84.3) | 0.577 (30.9) | 0.355 (43.9)
  M2 (BAY75-7495) (n=3,6,5,3,6,10,2,16) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 0.0855 (161) | 0.124 (37.0) | 0.169 (71.5) | 0.135 (20.3) | 0.148 (69.9) | 0.263 (74.6) | 0.113 (77.8)
  M5 (BAY81-8752) (n=3,8,10,6,10,1,4,24) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 0.0157 (NA) — we have one data point only, n=1, calculation not possible | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations)

8. Secondary Outcome: Maximum Observed Plasma Concentration After Single Dose Administration Divided by Dose (Cmax/D)
Description: Cmax/D refers to the highest measured drug concentration after a single dose administration, which is then divided by the administered dose. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 2
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmax/D in at least one analyte was 1 (M5) in 20mg; 7 (regorafenib and M2) and 5 (M5) in 40mg; 13 (M5) in HCC Child-Pugh A; 22 (M5) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
1/L
  Regorafenib (n=3,7,10,6,10,14,4,24) | 0.0165 (14.8) | 0.0106 (27.4) | 0.0125 (30.7) | 0.0156 (24.0) | 0.0136 (51.2) | 0.0138 (97.9) | 0.0142 (76.1) | 0.0125 (68.5)
  M2 (BAY75-7495) (n=3,7,10,6,10,14,4,24) | 0.000874 (244) | 0.00210 (110) | 0.00388 (51.2) | 0.00520 (43.2) | 0.00419 (97.2) | 0.00404 (154) | 0.00526 (129) | 0.00376 (190)
  M5 (BAY81-8752) (n=1,5,10,6,10,13,4,22) | 0.000114 (NA) — we have one data point only, n=1, calculation not possible | 0.000184 (124) | 0.000298 (118) | 0.000381 (59.2) | 0.000355 (140) | 0.000355 (110) | 0.000351 (352) | 0.000320 (142)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 2
Population: Pharmacokinetic population; Number of Participants with an evaluable Tmax in at least one analyte were 1 (M-5) in 20 mg; 5 (M-5) in 40mg; 13 (M-5) in HCC Child Pugh A; 22 (M-5) in NSCLC
Measure: Median (Full Range); unit: h
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
h
  Regorafenib (n=3,8,10,6,10,14,4,24) | 8.00 [4.00 to 34.0] | 2.02 [2.00 to 10.0] | 5.00 [2.00 to 48.0] | 6.00 [2.00 to 24.0] | 3.01 [1.00 to 24.7] | 3.03 [2.00 to 24.0] | 3.00 [2.00 to 10.0] | 2.00 [1.00 to 48.1]
  M2 (BAY75-7495) (n=3,8,10,6,10,14,4,24) | 8.00 [4.00 to 24.6] | 2.02 [2.00 to 10.0] | 10.0 [2.00 to 48.0] | 9.00 [2.00 to 24.0] | 4.00 [2.00 to 24.7] | 3.01 [2.00 to 24.0] | 10.0 [8.00 to 24.1] | 2.01 [2.00 to 48.0]
  M5 (BAY81-8752) (n=1,5,10,6,10,13,4,22) | 48.0 [48.0 to 48.0] | 47.8 [10.0 to 48.0] | 48.0 [24.0 to 48.0] | 24.6 [10.0 to 48.0] | 47.6 [24.1 to 48.0] | 46.8 [4.00 to 48.6] | 34.9 [24.0 to 46.8] | 47.8 [4.00 to 48.4]

10. Secondary Outcome: Half-life Associated With the Terminal Slope (T1/2)
Description: T1/2 is the period of time required for the concentration or amount of drug in the body to be reduced to exactly one-half of a given concentration or amount. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 2
Population: PK population; Number of Patients with at least an evaluable T1/2 were 5 (regorafenib) and 6 (M2) in 40mg; 5 (regorafenib and M2) in 100 mg; 3 (regorafenib and M2) in 120 mg; 6 (regorafenib and M2) in 140 mg; 9 (regorafenib), 10(M2) and 1 (M5) in HCC Child Pugh A; 3 (regorafenib) and 2 (M2) in HCC Child Pugh B; 19 (regorafenib) and 16 (M2) in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
h
  Regorafenib (n=3,5,5,3,6,9,22,19) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 41.6 (41.1) | 31.6 (32.5) | 27.7 (47.8) | 23.2 (43.6) | 25.2 (52.0) | 745.3 (79.7) | 33.3 (64.8)
  M2 (BAY75-7495) (n=3,6,5,3,6,10,2,16) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 40.3 (52.3) | 24.8 (28.6) | 22.9 (27.6) | 22.7 (64.7) | 24.0 (56.3) | 19.2 (16.4) | 26.4 (73.4)
  M5 (BAY81-8752) (n=3,8,10,6,10,1,4,24) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | 68.7 (NA) — we have one data point only, n=1, calculation not possible | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations) | NA (NA) — not calculated due to no evaluable data (i.e. insufficient plasma concentrations)

11. Secondary Outcome: Cmax at Steady State During a Dosing Interval Divided by Dose (Cmax,ss/D)
Description: Cmax,ss/D refers to the highest measured drug concentration after multiple dose administration and after a steady state concentration has been reached, which is then divided by the administered dose. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 4
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmax,ss/D in at least one analyte were 6 in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
1/L
  Regorafenib (n=3,6,6,2,3,0,1,5) | 0.0636 (19.4) | 0.0374 (37.0) | 0.0427 (22.9) | 0.0302 (5.77) | 0.0383 (30.9) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.0269 (NA) — we have one data point only, n=1, calculation not possible | 0.0255 (92.4)
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 0.00441 (39.5) | 0.0126 (74.3) | 0.0241 (36.3) | 0.0240 (217) | 0.0152 (106) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.0232 (NA) — we have one data point only, n=1, calculation not possible | 0.00881 (126)
  M5 (BAY81-8752) (n=3,6,6,2,3,0,1,5) | 0.000454 (15.7) | 0.00434 (151) | 0.0137 (87.9) | 0.0273 (1400) | 0.00674 (343) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.0159 (NA) — we have one data point only, n=1, calculation not possible | 0.00347 (153)

12. Secondary Outcome: AUC From Time 0 to 24 Hours at Steady State Divided by Dose (AUC(0-24)ss/D)
Description: AUC(0-24)ss/D is a measure of systemic drug exposure (AUC) over 24 hours after multiple dose administration and after a steady state concentration has been reached, which is then divided by the administered dose. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 5
Population: Pharmacokinetic population; Number of Participants with an evaluable AUC(0-24)ss/D in at least one analyte were 6 in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h/L
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
h/L
  Regorafenib (n=3,6,6,2,3,0,1,5) | 0.644 (21.2) | 0.452 (35.9) | 0.496 (18.5) | 0.338 (32.9) | 0.431 (18.5) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.392 (NA) — we have one data point only, n=1, calculation not possible | 0.358 (83.8)
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 0.0538 (42.9) | 0.174 (56.7) | 0.305 (25.2) | 0.330 (245) | 0.205 (88.8) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.453 (NA) — we have one data point only, n=1, calculation not possible | 0.141 (104)
  M5 (BAY81-8752) (n=3,6,6,2,3,0,1,5) | 0.00609 (18.7) | 0.0552 (136) | 0.185 (58.1) | 0.368 (3050) | 0.0916 (231) | NA (NA) — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.342 (NA) — we have one data point only, n=1, calculation not possible | 0.0615 (133)

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax,ss)
Description: Tmax,ss refers to the time after multiple dose administration and after a steady state concentration has been reached when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 5
Population: Pharmacokinetic population; Number of Participants with an evaluable Tmax,ss in at least one analyte were 6 in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Median (Full Range); unit: h
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
h
  Regorafenib (n=3,6,6,2,3,0,1,5) | 2.00 [2.00 to 4.00] | 2.00 [1.00 to 10.0] | 1.25 [0.00 to 4.00] | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 4.00] | NA [NA to NA] — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 4.03 [4.03 to 4.03] | 4.00 [2.00 to 10.0]
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 2.00 [2.00 to 4.00] | 1.50 [1.00 to 10.0] | 2.00 [0.00 to 8.00] | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 8.00] | NA [NA to NA] — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 10.0 [10.0 to 10.0] | 4.00 [2.00 to 10.0]
  M5 (BAY81-8752) (n=3,6,6,2,3,0,1,5) | 2.00 [0.500 to 4.00] | 1.00 [1.00 to 1.00] | 1.00 [0.00 to 24.0] | 1.50 [1.00 to 2.00] | 1.00 [0.00 to 8.00] | NA [NA to NA] — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.00 [0.00 to 0.00] | 4.00 [0.00 to 10.0]

14. Secondary Outcome: Ratio of Cmax,ss/Cmax (RACmax)
Description: RACmax is the ratio of the highest drug concentration at steady state to the highest drug concentration after single dose administration. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: Blood samples were collected on Cycle 1, Day 1 and Cycle 2, Day 1 and on Cycle 3, Day 1 for expansion cohort. Samples were drawn at the following time points: 0 h pre-dose, 0.5, 1, 2, 4, 8, 10 and 24h post-dose
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmax,ss and Cmax in at least one analyte were 1 (M5) in 20mg; 5 (regorafenib and M2) and 4 (M5) in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Number; unit: Ratio
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
Ratio
  Regorafenib (n=3,5,6,2,3,0,1,5) | 3.78 | 3.34 | 3.50 | 1.53 | 2.84 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 1.90 | 1.82
  M2 (BAY75-7495) (n=3,5,6,2,3,0,1,5) | 4.86 | 4.26 | 5.39 | 3.06 | 3.33 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 3.40 | 1.83
  M5 (BAY81-8752) (n=1,4,6,2,3,0,1,5) | 3.80 | 22.8 | 32.5 | 39.3 | 18.9 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 45.0 | 11.9

15. Secondary Outcome: Ratio of Cmin,ss/Cmin (RACmin)
Description: RACmin is the ratio of the lowest drug concentration at steady state to the lowest drug concentration after single dose administration. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 14
Population: Pharmacokinetic population; Number of Participants with an evaluable Cmin,ss and Cmin in at least one analyte were 0 (M5) in 20mg; 6 (regorafenib and M2) and 4 (M5) in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Number; unit: Ratio
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
Ratio
  Regorafenib (n=3,6,6,2,3,0,1,5) | 4.82 | 34.9 | 26.1 | 413 | 10.9 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 7.80 | 14.1
  M2 (BAY75-7495) (n=3,6,6,2,3,0,1,5) | 4.81 | 10.4 | 24.2 | 12.6 | 3.33 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 103 | 11.5
  M5 (BAY81-8752) (n=0,4,,6,2,3,0,1,5) | NA — 3 participants were analyzed. Not calculated due to no participant with an evaluable data | 26.1 | 102 | 335 | 46.2 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 257 | 22.4

16. Secondary Outcome: Ratio of AUCt,ss/AUCt (RAAUC)
Description: RAAUC is the ratio of the measure of systemic drug exposure over a specific dosing interval at steady state to the measure of systemic drug exposure over a specific dosing interval after single dose administration. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: as for outcome 14
Population: Pharmacokinetic population; Number of Participants with an evaluable AUCt,ss and AUCt in at least one analyte were 0 (M5) in 20mg; 5 (regorafenib and M2) and 4 (M5) in 40mg; 6 in 100 mg; 2 in 120 mg; 3 in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 5 in NSCLC
Measure: Number; unit: Ratio
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
Ratio
  Regorafenib (n=3,5,6,2,3,0,1,5) | 3.20 | 3.78 | 3.15 | 1.37 | 3.61 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 2.10 | 2.67
  M2 (BAY75-7495) (n=3,5,6,2,3,0,1,5) | 5.79 | 4.72 | 4.63 | 2.71 | 3.60 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 4.60 | 2.74
  M5 (BAY81-8752) (n=0,4,,6,2,3,0,1,5) | NA — 3 participants were analyzed. Not calculated due to no participant with an evaluable data | 28.1 | 41.2 | 34.7 | 23.9 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 63.0 | 18.5

17. Secondary Outcome: Ratio of AUCt,ss/AUC (RLIN)
Description: RLIN is the ratio of the measure of systemic drug exposure at steady state to the measure of systemic drug exposure after single dose administration. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: Blood samples were collected on Cycle 1, Day 1 and Cycle 2, Day 1. Samples were drawn at the following time points: 0 h pre-dose, 0.5, 1, 2, 4, 8, 10 and 24h post-dose
Population: PK population; Number of Participants with an evaluable AUCt,ss and AUC in at least one analyte were 0 in 20mg; 3 (regorafenib) and 4 (M2) in 40mg; 3 in 100 mg; 2 (regorafenib) and 0 (M2) in 120 mg; 3 (regorafenib) and 2 (M2) in 140 mg; 0 in HCC Child Pugh A; 1 in HCC Child Pugh B; 4 in NSCLC; No participants have evaluable data for M5.
Measure: Number; unit: Ratio
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg | HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg | HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 10 | 14 | 4 | 24
Ratio
  Regorafenib (n=0,3,3,2,3,0,1,4) | NA — 3 participants were analyzed. Not calculated due to no participant with an evaluable data | 1.53 | 1.27 | 0.600 | 2.20 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 0.800 | 1.11
  M2 (BAY75-7495) (n=0,4,3,0,2,0,1,4) | NA — 3 participants were analyzed. Not calculated due to no participant with an evaluable data | 1.63 | 2.13 | NA — 6 participants were analyzed. Not calculated due to no participant with an evaluable data | 1.39 | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | 2.70 | 1.27
  M5 (BAY81-8752) (n=0) | NA — 3 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 8 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 10 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 6 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 10 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 14 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 4 participants were analyzed. Not calculated due to no participant with an evaluable data | NA — 24 participants were analyzed. Not calculated due to no participant with an evaluable data

18. Secondary Outcome: Biomarker Vascular Endothelial Growth Factor (VEGF) Plasma Levels
Description: The analysis of Biomarker VEGF plasma levels is not done
Time Frame: No data obtained
Population: ITT
Arm/Group | Regorafenib, 20 mg, 40 mg, 100 mg, 120 mg, 140 mg
Number analyzed (Participants) | 0

19. Secondary Outcome: Biomarker Soluble Vascular Endothelial Growth Factor Receptor 2 (sCEGFR-2) Plasma Levels
Description: The analysis of Biomarker sCEGFR-2 plasma levels is not done.
Time Frame: No data obtained
Population: ITT
Arm/Group | Regorafenib, 20 mg, 40 mg, 100 mg, 120 mg, 140 mg
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Tumor Progression in Dose Escalation Cohort
Description: Tumor progression evaluates changes in a tumor or tumors over time due to worsening of disease. Measurements and observations of the tumor status were performed before, during and after treatment. Progression for solid tumors was evaluated based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.0) criteria. Tumor dimensions were measured in millimeters and the longest diameter (LD) was recorded for up to 5 lesions per organ and 10 lesions total. A sum of the LD for all target lesions was recorded. The use of a 20% increase in the sum of LD of target lesions from the smallest sum or appearance of a new lesion was assessed as progression of disease.
Time Frame: From the screening visit of the first participant until the last evaluation of the final participant over 6 years later, assessed at the screening visit, end of cycle 2, end of each even cycle and during the final visit (end of treatment)
Population: Intent-to-treat (ITT) efficacy analysis (set)
Measure: Number; unit: Participants
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg
Number analyzed (Participants) | 3 | 8 | 11 | 5 | 10
Participants
  Participants without progression | 1 | 3 | 9 | 2 | 5
  Participants with progression | 2 | 5 | 2 | 3 | 5

21. Other Pre Specified Outcome: Tumor Progression in Expansion Cohort
Description: Tumor progression evaluates changes in a tumor or tumors over time due to worsening of disease. Measurements and observations of the tumor status were performed before, during and after treatment. Tumor progression evaluates changes in a tumor or tumors over time due to worsening of disease. Measurements and observations of the tumor status were performed before, during and after treatment. Progression for solid tumors was evaluated based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.0) criteria. Tumor dimensions were measured in millimeters and the longest diameter (LD) was recorded for up to 5 lesions per organ and 10 lesions total. A sum of the LD for all target lesions was recorded. The use of a 20% increase in the sum of LD of target lesions from the smallest sum or appearance of a new lesion was assessed as progression of disease.
Time Frame: as for outcome 20
Population: ITT efficacy analysis (set), expansion cohorts only
Measure: Number; unit: Participants
Groups:
- HCC Expansion Cohort: Regorafenib 100 mg: Hepatocellular carcinoma (HCC) Participants with Child Pugh A or B status in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
Arm/Group | HCC Expansion Cohort: Regorafenib 100 mg | NSCLC Expansion Cohort: Regorafenib 100 mg
Number analyzed (Participants) | 22 | 22
Participants
  Participants without progression | 10 | 6
  Participants with progression | 12 | 16

22. Other Pre Specified Outcome: Tumor Response in Dose Escalation Cohort
Description: Tumor Response (= Best Overall Response) of a participant was defined as the best tumor response (Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes, SD was defined as steady state of disease, PD was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: as for outcome 20
Population: ITT efficacy analysis (set)
Measure: Number; unit: Participants
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg
Number analyzed (Participants) | 3 | 8 | 11 | 5 | 10
Participants
  Not assessable | 0 | 1 | 2 | 0 | 0
  Partial Response (PR) | 0 | 0 | 2 | 0 | 1
  Stable Disease (SD) | 1 | 2 | 5 | 2 | 4
  Progressive Disease (PD) | 2 | 4 | 2 | 2 | 4
  Progression | 0 | 1 | 0 | 1 | 1

23. Other Pre Specified Outcome: Tumor Response in Expansion Cohort
Description: as for outcome 22
Time Frame: as for outcome 20
Population: ITT efficacy analysis (set), expansion cohorts only
Measure: Number; unit: Participants
Groups:
- HCC Expansion Cohort, Regorafenib 100 mg: Hepatocellular carcinoma (HCC) Participants with Child Pugh A or B status in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
- NSCLC Expansion Cohort, Regorafenib 100 mg: Non-small cell lung cancer (NSCLC) participants in the expansion cohort received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets of regorafenib was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle.
Arm/Group | HCC Expansion Cohort, Regorafenib 100 mg | NSCLC Expansion Cohort, Regorafenib 100 mg
Number analyzed (Participants) | 22 | 22
Participants
  Not assessable | 3 | 1
  Partial Response (PR) | 1 | 0
  Stable Disease (SD) | 6 | 5
  Progressive Disease (PD) | 10 | 12
  Progression | 2 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected after signing the informed consent of the first participant until the end of study completion for the last patient, therefore for the study over a period of approximately 6 years and 9 months
Groups:
- Regorafenib (Stivarga, BAY73-4506) 100 mg: Participants received a single 100 mg oral CP tablet of regorafenib on Day 1 of Cycle 1 followed by 1 day off treatment. On Day 3, once-daily continuous dosing with 100 mg oral CP tablets was initiated. A cycle was defined as 21 days. For Cycle 2 and subsequent cycles, regorafenib was administered once daily continuously on a 21-day cycle. This arm includes the participants from the dose escalation cohort: Regorafenib 100 mg and the three Expansion Cohorts 'HCC Child-Pugh A Expansion Cohort: Regorafenib 100 mg', 'HCC Child-Pugh B Expansion Cohort: Regorafenib 100 mg', 'NSCLC Expansion Cohort: Regorafenib 100 mg'.
Arm/Group | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg | Regorafenib (Stivarga, BAY73-4506) 100 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/8 | 31/59 | 3/6 | 6/10
Other Adverse Events (participants affected / at risk) | 2/3 | 8/8 | 58/59 | 5/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg (N=3) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg (N=8) | Regorafenib (Stivarga, BAY73-4506) 100 mg (N=59) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg (N=6) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg (N=10)
Edema: Limb (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 0 | 0 | 3 | 0 | 2
Conduction abnormality, AV Block - 3rd Degree (Complete AV Block) (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
SupraVentricular arrhythmia, Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular - Other (Eye disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
GI - Other (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Obstruction, GI, Duodenum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Constitutional Symptoms - Other (General disorders) | 0 | 0 | 1 | 0 | 0
Death not associated with CTCAE term, Disease Progression NOS (General disorders) | 0 | 0 | 5 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 4 | 1 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 1
Pain, Abdomen NOS (General disorders) | 0 | 0 | 1 | 0 | 0
Pain, Back (General disorders) | 0 | 0 | 2 | 0 | 0
Pain, Chest wall (General disorders) | 0 | 0 | 1 | 0 | 0
Pain, Chest/thorax NOS (General disorders) | 0 | 1 | 0 | 1 | 0
Pain, Joint (General disorders) | 0 | 0 | 1 | 0 | 0
Pain, Other (Specify) (General disorders) | 0 | 0 | 1 | 0 | 0
Liver dysfunction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Infection (Documented clinically), Appendix (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Infection (Documented clinically), Blood (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Documented clinically), Bronchus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Documented clinically), Lung (pneumonia) (Infections and infestations) | 0 | 0 | 4 | 1 | 0
Infection (Documented clinically), Urinary tract NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection with normal ANC, Colon (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Secondary Malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Renal - Other (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
CNS hemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hemorrhage pulmonary, Respiratory tract NOS (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 20 mg (N=3) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 40 mg (N=8) | Regorafenib (Stivarga, BAY73-4506) 100 mg (N=59) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 120 mg (N=6) | Escalation Cohort: Regorafenib (Stivarga, BAY73-4506) 140 mg (N=10)
Blood - Other (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 0 | 1 | 11 | 2 | 3
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 5 | 1 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1
Platelets (Blood and lymphatic system disorders) | 0 | 1 | 9 | 1 | 0
Cardiac General - Other (Cardiac disorders) | 0 | 0 | 4 | 1 | 1
Hypertension (Cardiac disorders) | 0 | 0 | 21 | 2 | 2
Hypotension (Cardiac disorders) | 0 | 0 | 2 | 2 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1 | 0
SupraVentricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
SupraVentricular arrhythmia, Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
SupraVentricular arrhythmia, Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 3
Ventricular arrhythmia, Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 | 0 | 2 | 1 | 1
Hearing (without monitoring program) (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Otitis, external (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Hot flashes (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 13 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 2 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 0 | 22 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 14 | 3 | 3
Dehydration (Gastrointestinal disorders) | 0 | 0 | 7 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 15 | 2 | 4
Distension (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 8 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
GI - Other (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mucositis (clinical exam), Oral cavity (Gastrointestinal disorders) | 0 | 2 | 5 | 1 | 1
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 0 | 0 | 11 | 3 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 17 | 2 | 3
Taste Alteration (Gastrointestinal disorders) | 0 | 0 | 5 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 13 | 1 | 2
Constitutional Symptoms - Other (General disorders) | 1 | 1 | 2 | 1 | 1
Fatigue (General disorders) | 2 | 5 | 28 | 4 | 5
Fever (General disorders) | 0 | 0 | 9 | 1 | 2
Insomnia (General disorders) | 0 | 1 | 11 | 0 | 4
Pain, Abdomen NOS (General disorders) | 1 | 2 | 9 | 2 | 3
Pain, Anus (General disorders) | 0 | 0 | 0 | 1 | 0
Pain, Back (General disorders) | 0 | 1 | 13 | 4 | 2
Pain, Bladder (General disorders) | 0 | 0 | 0 | 1 | 0
Pain, Buttock (General disorders) | 0 | 0 | 3 | 0 | 0
Pain, Chest wall (General disorders) | 0 | 0 | 5 | 1 | 2
Pain, Chest/thorax NOS (General disorders) | 0 | 0 | 3 | 1 | 0
Pain, Dental/teeth/peridontal (General disorders) | 0 | 0 | 1 | 0 | 1
Pain, Extremity - limb (General disorders) | 0 | 0 | 15 | 5 | 5
Pain, Head/headache (General disorders) | 0 | 1 | 8 | 2 | 1
Pain, Joint (General disorders) | 0 | 1 | 6 | 2 | 1
Pain, Muscle (General disorders) | 0 | 0 | 10 | 4 | 3
Pain, Neuralgia/peripheral nerve (General disorders) | 0 | 0 | 1 | 1 | 0
Pain, Oral cavity (General disorders) | 0 | 0 | 1 | 0 | 1
Pain, Other (Specify) (General disorders) | 1 | 1 | 4 | 1 | 3
Pain, Pain NOS (General disorders) | 0 | 0 | 7 | 0 | 0
Pain, Scalp (General disorders) | 0 | 0 | 0 | 1 | 0
Pain, Throat/pharynx/larynx (General disorders) | 0 | 0 | 5 | 0 | 0
Pain, Tumor pain (General disorders) | 0 | 2 | 1 | 0 | 2
Rigors/chills (General disorders) | 0 | 0 | 3 | 1 | 2
Sweating (General disorders) | 0 | 1 | 6 | 1 | 1
Syndromes - Other (General disorders) | 0 | 0 | 0 | 0 | 1
Weight loss (General disorders) | 0 | 0 | 2 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Allergy - Other (Immune system disorders) | 0 | 1 | 1 | 0 | 2
Rhinitis (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Infection (Documented clinically), Abdomen NOS (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Infection (Documented clinically), Bronchus (Infections and infestations) | 0 | 1 | 4 | 0 | 0
Infection (Documented clinically), Conjunctiva (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Documented clinically), Lip/perioral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Documented clinically), Neck NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Documented clinically), Pharynx (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Infection (Documented clinically), Upper airway NOS (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Infection (Documented clinically), Urinary tract NOS (Infections and infestations) | 0 | 0 | 5 | 1 | 1
Infection - Other (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Infection with normal ANC, Anal/perianal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection with normal ANC, Pharynx (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Infection with normal ANC, Sinus (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 0 | 0 | 3 | 1 | 1
ALT (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1
AST (Metabolism and nutrition disorders) | 0 | 0 | 7 | 0 | 2
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 7 | 0 | 5
CPK (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Cholesterol (serum-high hypercholesteremia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 6 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 8 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 10 | 2 | 2
Lipase (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 0 | 1 | 5 | 1 | 2
Proteinuria (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Gait/walking (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 2 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 1
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 0 | 3 | 9 | 0 | 0
Secondary Malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
CNS ischemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 6 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Mood Alteration, Agitation (Nervous system disorders) | 1 | 0 | 1 | 1 | 1
Mood Alteration, Anxiety (Nervous system disorders) | 0 | 0 | 5 | 2 | 3
Mood Alteration, Depression (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Neurology - Other (Nervous system disorders) | 0 | 1 | 3 | 0 | 1
Neuropathy: Cranial, CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Neuropathy: Cranial, CN XI Motor-Sternomastoid And Trapezius (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy: Cranial, CN XII Motor-tongue (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Neuropathy: sensory (Nervous system disorders) | 0 | 2 | 13 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Renal - Other (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 18 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 14 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 9 | 2 | 2
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 13 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 1 | 2
Bruising (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Burn (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis, Radiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 | 2 | 10 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 9 | 1 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 23 | 2 | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 6 | 19 | 5 | 9
Hemorrhage pulmonary, Nose (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Hemorrhage, GI, Anus (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vascular - Other (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No